CLINICAL TRIAL: NCT05687305
Title: The Effect of White Noise on Sleep Quality, Comfort and Satisfaction Level in Patients Undergoing Lumbar Disc Herniation Surgery: A Randomized Controlled Study
Brief Title: The Effect of White Noise in Patients Undergoing Lumbar Disc Herniation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 27.05.2022-22-36
Record Dates: First submitted 2022-12-30; First posted 2023-01-18 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Disc Herniation
Keywords: Lumbar Disc Herniation; White Noise; Sleep Quality; Comfort Level
MeSH Terms: conditions — Intervertebral Disc Displacement; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is a single-center parallel-group randomized controlled clinical trial.
  Participants who accepted to participate in the study and met the inclusion criteria will be assigned to the intervention (n=30) or control group (n=30) according to the computer-based randomization table.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): On the 0th and 1st postoperative days, patients in the intervention group will listen to white noise with a bluetooth headset for 30 minutes before going to sleep, and they will be kept under observation during this time.Patients in the control group will be monitored according to their routine clinical procedures. Since there are no procedures or interventions in clinical procedures, only patient monitoring will be performed. Patients in the control group will also be followed up at the same times and with the same forms.
  Interventions: Other: White Noise
- No Intervention Group (No Intervention): Patients in the control group will not receive any intervention other than their routine. Data collection forms will be applied to the participants in the control group at the same time as the intervention group.

INTERVENTIONS:
Other: White Noise — White noise is produced by digitally combining sounds of equal frequency in the laboratory. Then, all of the frequencies in this sound are calibrated to generate noise at each frequency. If the contribution of each region to the noise level is the same, the noise is referred to as white noise. Waterfalls, ocean waves, and wind blowing through trees all produce similar to white noise. Patients in the intervention group are observed by the investigator on the 0th and 1st postoperative days.Before going to sleep, a bluetooth headset will be used to listen to white noise for 30 minutes and vital signs will be measured before and after the procedure.
  Arms: Intervention Group

SUMMARY:
The aim of this clinical trial is to determine the effectiveness of listening to white noise on the sleep quality, comfort level, satisfaction level of patients after lumbar disc herniation surgery. The main hypotheses are:

* Is there a difference between the sleep quality of patients who listen to white noise and those who do not?
* Is there a difference between the comfort levels of patients who listen to white noise and those who do not?
* Is there a difference between the satisfaction levels of patients who listen to white noise and those who do not?

The main tasks that the participants will be asked to do will be explained and Their informed consent will be obtained. The two research groups will be compared.

DETAILED DESCRIPTION:
This study will be conducted with a total of 60 patients who underwent surgery for lumbar disc herniation at a hospital in Istanbul. Participants in the study who had lumbar disc herniation surgery will be divided into two groups: intervention (n = 30) and control group (n = 30), according to the randomization method created with computer-based random numbers.

On the 0th and 1st postoperative days, patients in the intervention group will listen to white noise with a bluetooth headset for 30 minutes before going to sleep, and they will be kept under observation during this time.Patients in the control group will be monitored according to their routine clinical procedures. Since there are no procedures or interventions in clinical procedures, only patient monitoring will be performed. Patients in the control group will also be followed up at the same times and with the same forms. Descriptive Characteristics Form, Informed Consent Form, The Richards-Campbell Sleep Questionnaire, General Comfort Questionnaire,Visual Analog Scale for Satisfaction Level will be used in data collection.

ELIGIBILITY:
Inclusion Criteria:

* underwent lumbar disc herniation surgery
* hospitalized for at least 48 hours
* agreed to participate in research

Exclusion Criteria:

* chronic sleep problems and taking medication
* Not filling out the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change of Sleep Quality Assessed by the Richard Campbell Sleep Scale | Change from baseline sleep quality at two days after surgery
  The sleep quality of the patients was evaluated with the Richard Campbell Sleep Scale on the 1st and 2nd postoperative days after morning treatment. This scale consists of 6 items and the total score range is 0-100 points. As the scale score increases, the sleep quality of the patients also increases.
Change of Comfort Level Assessed by the General Comfort Questionnaire Short Form | Change from baseline comfort level at two days after surgery
  The general comfort levels of the patients were evaluated with the General Comfort Questionnaire Short Form after the morning treatment on the 1st and 2nd postoperative days. This scale consists of 28 items and includes three sub-dimensions; comfort, relaxation and relaxation. The scale score is calculated by dividing the total score obtained from the scale by the number of scale items. The scale total score range is between 0-6 points. As the scale score increases, the comfort level of the patients also increases.
Change of Satisfaction Level Assessed by Visual Analogue Scale | Change from baseline satisfaction level at two days after surgery
  The satisfaction levels of the patients were evaluated with the Visual Analogue Scale on the 1st and 2nd postoperative days, after the morning treatment. This scale consists of 10 cm horizontal lines and is evaluated between 0-10 points. As the scale score increases, the satisfaction level of the patients also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Kızılkaya, RN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Melike Kızılkaya, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murase K, Tabara Y, Ito H, Kobayashi M, Takahashi Y, Setoh K, Kawaguchi T, Muro S, Kadotani H, Kosugi S, Sekine A, Yamada R, Nakayama T, Mishima M, Matsuda S, Matsuda F, Chin K. Knee Pain and Low Back Pain Additively Disturb Sleep in the General Population: A Cross-Sectional Analysis of the Nagahama Study. PLoS One. 2015 Oct 7;10(10):e0140058. doi: 10.1371/journal.pone.0140058. eCollection 2015. PMID 26444713
- [Result] Chou R, Baisden J, Carragee EJ, Resnick DK, Shaffer WO, Loeser JD. Surgery for low back pain: a review of the evidence for an American Pain Society Clinical Practice Guideline. Spine (Phila Pa 1976). 2009 May 1;34(10):1094-109. doi: 10.1097/BRS.0b013e3181a105fc. PMID 19363455
- [Result] Kavcic N, Grenier S, McGill SM. Quantifying tissue loads and spine stability while performing commonly prescribed low back stabilization exercises. Spine (Phila Pa 1976). 2004 Oct 15;29(20):2319-29. doi: 10.1097/01.brs.0000142222.62203.67. PMID 15480148
- [Result] Akiyama A, Tsai JD, W Y Tam E, Kamino D, Hahn C, Go CY, Chau V, Whyte H, Wilson D, McNair C, Papaioannou V, Hugh SC, Papsin BC, Nishijima S, Yamazaki T, Miller SP, Ochi A. The Effect of Music and White Noise on Electroencephalographic (EEG) Functional Connectivity in Neonates in the Neonatal Intensive Care Unit. J Child Neurol. 2021 Jan;36(1):38-47. doi: 10.1177/0883073820947894. Epub 2020 Aug 24. PMID 32838628